CLINICAL TRIAL: NCT04221516
Title: Camrelizumab After Completion of Radiotherapy for Oligometastatic Nasopharyngeal Carcinoma: A Phase 2 Trial
Brief Title: Camrelizumab After Completion of Radiotherapy for Oligometastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2019-184
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Carcinoma; Oligometastasis; Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab (Experimental): Camrelizumab 200mg every 21 days for up to 18 cycles, from 4 to 12 weeks after the completion of radiotherapy.
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg every 21 days (3 weeks) for up to 18 cycles, from 4 to 12 weeks after the completion of radiotherapy.

SUMMARY:
The main purpose of this study is to see how well the experimental drug camrelizumab(SHR-1210) works in people with oligometastatic NPC who have already had locally radiotherapy for their disease. All patients will receive 200 mg of camrelizumab intravenously on Day 1 of each 21-day cycle. Patients will receive the study drug for up to 18 cycles.

DETAILED DESCRIPTION:
Each subject included in this project must sign an informed consent form. Within 4-6 weeks after completing radiotherapy and chemotherapy for oligometastatic lesions, subjects will receive camrelizumab 200 mg fixed-dose treatment every three-week (Q3W).

If there is no confirmed disease progression, unacceptable adverse events or concurrent diseases (need further treatment ), the researcher decides to withdraw from the subject, the subject withdraws from treatment, the subject is pregnant, and other reasons that do not meet the requirements of the trial treatment or procedure, The treatment with camrelizumab will last at least 12 months. Patients with no signs of disease progression can be treated with another 6 to 12 months by the decision of researcher.

After treatment, each subject will be followed up. Subjects should be monitored for adverse events for at least 30 days, and serious adverse events will be over 90 days. Subjects will be followed up 5 years from the last treatment or until one of the following events: ① disease progression; ② receive other treatments of cancer; ③ withdraw research consent; ④ loss of follow-up; ⑤ death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed non-keratinizing (according to World Health Organization (WHO) histologically type).
* Patients with oligometastatic NPC (defined as ≤5 metastases, ≤2 organs), without local recurrence of nasopharynx.
* Completion of radiotherapy 4-12 weeks prior to enrollment. At list one cycle of adjuvant platinum-based chemotherapy.
* Satisfactory performance status: Karnofsky scale (KPS) > 70.
* Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.
* Adequate renal function: creatinine clearance ≥50 ml/min.
* Expected lifetime over 3 months
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* Previous history of autoimmune disease or unstable autoimmune disease.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections are not excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome are not excluded from the study.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 3 years
  Time to progression or death from initiation of Camrelizumab
Drug toxicity and tolerability | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Life Quality | 3 years
  Evaluate patient quality of life by EORTC QLQ-C30 scale(Scores range from 0 to 100,a high functional scale score represents a high/healthy level of functioning, while a high symptom scale score indicates a high level of symptomatology or problems)
Overall Survival | 3 years
  Time to death from initiation of Camrelizumab

OTHER OUTCOMES:
Potential predictive biomarkers associated with therapeutic efficacy and prognosis | 3 years
  PD-L1 expression;Tumor Mutational Burden(TMB);Tumor related gene changes; plasma EBV DNA copies ; cytokine; etc

CONTACTS AND LOCATIONS:
Overall Officials: Jian Guan, Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Southern medical university, Guangzhou, Guangdong, China